CLINICAL TRIAL: NCT02880735
Title: Effect of Noninvasive Mechanical Ventilation on Ventilatory Response in Patients With Myotonic Dystrophy Type 1
Brief Title: Ventilatory Response After Non Invasive Ventilation in Type 1 Myotonic Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C46-15
Record Dates: First submitted 2016-08-12; First posted 2016-08-26 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Myotonic Dystrophy 1; Steinert Disease
Keywords: Myotonic Dystrophy; Noninvasive Ventilation; Respiratory Failure
MeSH Terms: conditions — Myotonic Dystrophy; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non Invasive Ventilation. (Experimental): It will provide noninvasive mechanical ventilation with the following specifications:
  Bilevel devices: Pressurized bilevel mode Spontaneous/Time. Interface: Facial mask Usage: During sleep Frequency: Daily Duration: Three months.
  Interventions: Device: Non Invasive Ventilation.

INTERVENTIONS:
Device: Non Invasive Ventilation. — Non Invasive Mechanical Ventilation through oronasal mask. Mode: Bilevel with rate backup (spontaneous/time). Inspiratory Pressure: 30-10, Expiratory Pressure : 4-15, Backup Rate;14-25 rpm. Use Time: During Sleep.

SUMMARY:
It has been suggested that patients with Myotonic Dystrophy type 1 have primary altered ventilatory response to chemical stimuli and chronic hypoventilation is related not always to muscle weakness. Also, it is known that Non Invasive Mechanical Ventilation can improve ventilatory response to chemical stimuli, especially to hypercapnia.

This study evaluates the effect of Non Invasive Mechanical Ventilation on ventilatory response in patients with Type 1 Myotonic Dystrophy, the ventilatory response to chemical stimuli will be measured before and after mechanical ventilation in patients with myotonic dystrophy type 1.

DETAILED DESCRIPTION:
Type 1 Myotonic Dystrophy is a hereditary neuromuscular disease with an autosomal dominant pattern whose prevalence is 1/8000 inhabitants and is the most common muscular dystrophy in adults. It is multisystem disease and is characterized by myotonia, progressive muscle loss and a wide spectrum of manifestations.

Myotonic dystrophy type 1 causes a high impact on health and quality of life of patients as functional impairment can reach the incapacity and total dependence in basic activities of daily living. As in most neuromuscular diseases, progressive muscle weakness at some point in the evolution affects the respiratory muscles. However, in some patients with myotonic dystrophy type 1 it has been observed that muscle weakness does not explain ventilatory failure, and is believed to be due to a primary reduction in the central ventilatory response to hypercapnia present in this disease.

Non Invasive Mechanical Ventilation (NIV) is a long-term treatment that provides ventilatory assistance through an interface that does not invade the airway and currently can be provided to patients in the home environment; It is a resource that has shown to improve the quality of life, daytime gas exchange and survival in patients with neuromuscular diseases, even when used only during sleep. It is not clear the mechanism by which NIV during daytime sleep improves gas exchange in patients with neuromuscular diseases, even in advanced stages where breathing muscles effectors are severely affected.

It has been proposed that NIV used during sleep can improve the sensitivity of the respiratory center to carbon dioxide but this has not been demonstrated in patients with Type 1 Myotonic Dystrophy, to answer this question, it is proposed to compare the central ventilatory response to chemical stimuli after a period of NIV in patients with Type 1 Myotonic Dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Classic variety of Myotonic Dystrophy Type 1
* Molecular confirmation through the standard method

Exclusion Criteria:

* Using currently invasive mechanical ventilation.
* Acute decompensation of respiratory or cardiac origin in the last 6 months, which required hospital care.
* Drugs that may alter the ventilatory response: benzodiazepines, neuroleptics, corticosteroids, theophylline, acetazolamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Ventilatory Response to Chemical Stimuli | Three months
  Increase the minute volume per unit of hypercapnia or hypoxemia, in a test of acute stimulation.

SECONDARY OUTCOMES:
Health Related Quality of Life Measured by Short Form 36 (SF-36) | Three months
  Scale for measuring the quality of life related to health in 8 domains (vitality, physical functioning, bodily pain, general health perception, physical role functioning, emotional role functioning, social role functioning, mental health), each rated from 0 to 100%. The higher score means better quality of life.
Dyspnoea evaluated by the modified scale of the Medical Research Council (mMRC) | Three months
  Rate dyspnea at 5 degrees from 0 to 5. 0: Not troubled by breathless except on strenuous exercise. 1: Short of breath when hurrying on a level or when walking up a slight hill. 2: Walks slower than most people on the level, stops after a mile or so, or stops after 15 minutes walking at own pace. 3: Stops for breath after walking 100 yards, or after a few minutes on level ground. 4: Too breathless to leave the house, or breathless when dressing/undressing.
Sleep Quality assessed by The Pittsburgh Sleep Quality Index (PSQI) | three months
  Assesses sleep quality. Contains 19 questions, each weighted on a 0-3 interval scale. A global PSQI score is taken from the survey, with lower scores correlating to better sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rogelio Perez Padilla, MD, Study Chair — National Institute of Respiratory Diseases, Mexico; Martha G Torres Fraga, MD, Principal Investigator — National Institute of Respiratory Diseases, Mexico
Locations (1):
- National Institute Of Respiratory Diseases, México, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Participant data to be shared will be: Results of functional testing and prescription ventilation.

REFERENCES:
- [Result] Meola G. Clinical aspects, molecular pathomechanisms and management of myotonic dystrophies. Acta Myol. 2013 Dec;32(3):154-65. PMID 24803843
- [Result] Mankodi A, Thornton CA. Myotonic syndromes. Curr Opin Neurol. 2002 Oct;15(5):545-52. doi: 10.1097/00019052-200210000-00005. PMID 12351998
- [Result] Carroll JE, Zwillich CW, Weil JV. Ventilatory response in myotonic dystrophy. Neurology. 1977 Dec;27(12):1125-8. doi: 10.1212/wnl.27.12.1125. PMID 563010
- [Result] Poussel M, Thil C, Kaminsky P, Mercy M, Gomez E, Chaouat A, Chabot F, Chenuel B. Lack of correlation between the ventilatory response to CO2 and lung function impairment in myotonic dystrophy patients: evidence for a dysregulation at central level. Neuromuscul Disord. 2015 May;25(5):403-8. doi: 10.1016/j.nmd.2015.02.006. Epub 2015 Feb 17. PMID 25753091
- [Result] Jammes Y, Pouget J, Grimaud C, Serratrice G. Pulmonary function and electromyographic study of respiratory muscles in myotonic dystrophy. Muscle Nerve. 1985 Sep;8(7):586-94. doi: 10.1002/mus.880080708. PMID 4047090
- [Result] Brooks D, De Rosie J, Mousseau M, Avendano M, Goldstein RS. Long term follow-up of ventilated patients with thoracic restrictive or neuromuscular disease. Can Respir J. 2002 Mar-Apr;9(2):99-106. doi: 10.1155/2002/545612. PMID 11972163
- [Result] Annane D, Quera-Salva MA, Lofaso F, Vercken JB, Lesieur O, Fromageot C, Clair B, Gajdos P, Raphael JC. Mechanisms underlying effects of nocturnal ventilation on daytime blood gases in neuromuscular diseases. Eur Respir J. 1999 Jan;13(1):157-62. doi: 10.1183/09031936.99.13115799. PMID 10836341